CLINICAL TRIAL: NCT01942083
Title: A Phase I, Open Label, Non Randomized, Multicenter, Dose Escalation Clinical Study to Investigate Safety and Tolerability of OPB(Otsuka Pharmaceutical Biwa)-111077 in Subjects With Advanced HCC(Hepatocellular Carcinoma)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company decision
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 317-12-001; There is no secondary ID.
Record Dates: First submitted 2013-06-26; First posted 2013-09-13 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Advanced Hepatocellular Carcinoma

STUDY DESIGN:
Intervention Model Description: Dose escalation study
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPB-111077 (Experimental): orally, once daily
  Interventions: Drug: OPB-111077

INTERVENTIONS:
Drug: OPB-111077

SUMMARY:
This is a Phase I, open label, non randomized, multicenter study designed to investigate the safety and tolerability of escalating doses of OPB-111077 administered orally, once daily in subjects with advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically or clinically diagnosed HCC by Korean Liver Cancer Study Group (KLCSG) guidelines.
2. Subject who has advanced HCC
3. Documented evidence of unresponsiveness to, intolerance to, or ineligibility for sorafenib, or unavailability of appropriate sorafenib treatment
4. Male or female subject, age at consent ≥20 years and ≤75 years.
5. Life expectancy ≥12 weeks.
6. Subjects who agree that they or their partner(s) will practice contraception during the study period and 3 months (12 weeks) after the completion of study treatment.
7. Subjects informed of the diagnosis of advanced HCC who are fully informed about the content of the study by the Investigator using the written consent form, and give written consent to participate in the study of their own free will.

Exclusion Criteria:

1. Past liver transplantation
2. Uncontrollable hepatic encephalopathy or ascites
3. Presence of brain metastases
4. Clinically significant gastrointestinal bleeding in past 6 months or current active gastrointestinal bleeding.
5. Primary malignancy other than HCC
6. Human immunodeficiency virus (HIV) infection
7. Severe or poorly controlled complication that may affect the conduct or results of the study.
8. Use of Interferon preparation within 4 weeks (28 days) before start of study treatment in the present study.
9. Pregnant, nursing, or possibly pregnant women, or women desiring to become pregnant during the study period
10. Other cases judged by the Investigator to be ineligible for participation in the study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-05-29 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-07-11 (Actual)

PRIMARY OUTCOMES:
Safety of OPB-111077 | Within the first cycle [24 days]
  Number of participants with adverse events as assessed by CTCAE v4.0
To investigate the maximum tolerated dose (MTD) of OPB-111077 | Within the first cycle [24 days]
  • The highest dose that does not lead to discontinuation of dose escalation is defined as the MTD.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) properties of OPB-111077 and its metabolites. | Within the first cycle [24 days]
  The following PK parameters (Cmax (maximum observed concentration), AUC(area uder the concentration time curve from zero), tmax (Time to maximum plasma concentration), etc.) will be determined using a non-compartmental methods.
Tumor response measured by RECIST(Response Evaluation Criteria in Solid Tumor) 1.1 | Approximately 3-18 weeks depending on tumor response
  Assessment will be conducted at Screening, end of Cycle 1, end of Cycle 2, end of every 2 cycles thereafter, at the Early Termination (discontinuation) Visit.
Biomarker of OPB-111077 | Within the first cycle [24 days]
  Change from baseline on predictable biomarker specified in the protocol

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul & Gyeonggi-Do, South Korea